CLINICAL TRIAL: NCT07126678
Title: Prospective Exploratory Study of Fixed-Duration Zanubrutinib, Bendamustine, and Obinutuzumab (ZBG) in Treatment-Naïve Advanced Stage Follicular Lymphoma
Brief Title: Fixed-Duration Zanubrutinib, Bendamustine, and Obinutuzumab (ZBG) in Treatment-Naïve Advanced Stage Follicular Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FL-ZBG-01
Record Dates: First submitted 2025-07-21; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Follicular Lymphoma; Treatment Naive
Keywords: Follicular lymphoma; fixed-duration; zanubrutinib; ZBG; Treatment Naive
MeSH Terms: conditions — Lymphoma, Follicular | interventions — zanubrutinib; Bendamustine Hydrochloride; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZBG (Experimental)
  Interventions: Drug: zanubrutinib, bendamustine, and obinutuzumab

INTERVENTIONS:
Drug: zanubrutinib, bendamustine, and obinutuzumab — Patients will receive combination therapy with zanubrutinib, bendamustine, and obinutuzumab over 6 cycles, with each cycle lasting 28 days. The specific dosing schedule is as follows: Bendamustine 70 mg/m²: administered intravenously on Days 2-3 of Cycle 1, and on Days 1-2 of Cycles 2-6. Obinutuzumab 1000 mg: administered intravenously on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-6 (every 28-day cycle). Zanubrutinib 160 mg orally twice daily (bid), continuously throughout Cycles 1-6.
  Treatment is discontinued after 6 cycles, with no subsequent maintenance therapy.

SUMMARY:
This study investigates a fixed-duration regimen of zanubrutinib, bendamustine, and obinutuzumab (ZBG) in the treatment of treatment-naïve patients with advanced-stage follicular lymphoma.

Patients will receive combination therapy with zanubrutinib, bendamustine, and obinutuzumab over 6 cycles, with each cycle lasting 28 days. The specific dosing schedule is as follows: Bendamustine 70 mg/m²: administered intravenously on Days 2-3 of Cycle 1, and on Days 1-2 of Cycles 2-6. Obinutuzumab 1000 mg: administered intravenously on Days 1, 8, and 15 of Cycle 1, and on Day 1 of Cycles 2-6 (every 28-day cycle). Zanubrutinib 160 mg orally twice daily (bid), continuously throughout Cycles 1-6.

Treatment is discontinued after 6 cycles, with no subsequent maintenance therapy.

Primary endpoint is 2-year PFS. Secondary endpoints include: CR rate after 6 cycles, ORR after 3 and 6 cycles MRD-negative rate after 3 and 6 cycles, OS, safety and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation with signed informed consent;
2. Age ≥18 years and ≤75 years, regardless of gender;
3. Life expectancy ≥3 months;
4. ECOG performance status 0-2; patients with ECOG 3 may be enrolled only if their decline in performance status is disease-related and the investigator judges they may benefit from treatment;
5. Histologically confirmed diagnosis of grade I, II, or IIIa follicular lymphoma (FL), treatment-naïve, stage III-IV disease, and meeting treatment criteria (GELF criteria);
6. Measurable and/or evaluable lymphoma lesions;
7. Adequate bone marrow reserve: absolute neutrophil count (ANC) >1.0×10⁹/L or platelets >75×10⁹/L, unless cytopenia is deemed related to bone marrow infiltration by lymphoma and the investigator believes it may recover;
8. Liver function: AST (SGOT), ALT (SGPT) ≤2.5×ULN (without liver involvement) or ≤5×ULN (with liver involvement); total bilirubin (TBIL) ≤ULN; serum creatinine (CRE) ≤1.5×ULN;
9. Creatinine clearance ≥30 mL/min (calculated by Cockcroft-Gault formula);
10. Ability to comply with study visit schedules and other protocol requirements;
11. All patients of childbearing potential must agree to use effective contraception during the study and for 24 months after treatment cessation; women of childbearing potential must have a negative urine pregnancy test before treatment initiation.

Exclusion Criteria:

1. Grade IIIb FL or transformed FL;
2. Received lymphoma-directed therapy within 2 weeks prior to enrollment;
3. Any severe medical condition, including but not limited to:

   * Poorly controlled hypertension (defined as failure to achieve control despite lifestyle modifications and treatment with at least 3 maximally tolerated antihypertensive drugs [including diuretics] for ≥4 weeks, or requiring ≥4 antihypertensive drugs for adequate control);
   * Uncontrolled congestive heart failure (NYHA class 3 [moderate] or 4 [severe]) within 6 months prior to screening;
   * Left ventricular ejection fraction (LVEF) <50%;
   * Symptomatic coronary artery disease (e.g., chest pain, palpitations, fatigue) or requiring medication;
   * Severe bradycardia (heart rate <40 bpm), hypotension, dizziness, or syncope; patients with arrhythmia history require cardiac evaluation;
   * Active bacterial, viral, fungal, or other infections (except for nail fungal infections) or major infections within 2 weeks before the first dose of study drug;
   * Moderate to severe liver disease (Child-Pugh B or C);
   * Active bleeding within 2 months before screening or clinically significant bleeding tendency per investigator judgment;
   * Pulmonary conditions impairing function (e.g., pulmonary fibrosis, drug-induced pneumonitis) deemed intolerable by the investigator;
   * Any psychiatric or cognitive impairment that may compromise understanding of informed consent, protocol compliance, or study adherence;
4. Known active hepatitis C virus (HCV) infection; other acquired/congenital immunodeficiency disorders, including HIV infection;
5. Central nervous system (CNS) involvement by lymphoma;
6. Diagnosis or treatment for malignancies other than lymphoma, except:

   * Malignancies treated with curative intent and no evidence of disease for ≥5 years before enrollment;
   * Adequately treated basal cell carcinoma (excluding melanoma) with no evidence of disease;
   * Adequately treated cervical carcinoma in situ with no evidence of disease;
7. Hypersensitivity to any study drug;
8. Pregnant or breastfeeding women;
9. History of stroke or intracranial hemorrhage within 6 months before enrollment;
10. Requiring anticoagulation with warfarin or equivalent vitamin K antagonists;
11. Requiring chronic use of strong CYP3A inhibitors;
12. Administration of live attenuated vaccines within 4 weeks before study entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year PFS | 2 year
  2-year progression-free survival (PFS)

SECONDARY OUTCOMES:
CR Rate | At the end of Cycle 6 (each cycle is 28 days)
  complete remission rate
ORR | At the end of Cycle 3 and 6 (each cycle is 28 days)
  objective remission rate
MRD | At the end of Cycle 6 (each cycle is 28 days)
  minimal residue rate
OS | From date of randomization until the date of death from any cause, assessed up to 100 months
  Overall survival
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE | 2 year
  * Adverse events and serious adverse events
  * Treatment-related adverse events leading to dose adjustments, dose interruptions, delays, and/or study drug discontinuation

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Serna A, Navarro V, Iacoboni G, Lopez L, Sancho JM, Gonzalez-Barca E, Lopez-Garcia A, Cordoba R, Saez A, Jimenez-Ubieto A, Ferrero A, Garcia T, Sanchez A, Garcia C, Bosch M, Cabirta A, Jimenez M, Marin-Niebla A, Bosch F, Abrisqueta P. Rituximab maintenance after bendamustine-based treatment for follicular lymphoma and mantle cell lymphoma may exert a negative influence on SARS-CoV-2 infection outcomes. Haematologica. 2025 Jan 1;110(1):173-178. doi: 10.3324/haematol.2024.285219. No abstract available. PMID 38988269
- [Background] Fowler NH, Nastoupil L, De Vos S, Knapp M, Flinn IW, Chen R, Advani RH, Bhatia S, Martin P, Mena R, Davis RE, Neelapu SS, Eckert K, Ping J, Co M, Beaupre DM, Neuenburg JK, Palomba ML. The combination of ibrutinib and rituximab demonstrates activity in first-line follicular lymphoma. Br J Haematol. 2020 May;189(4):650-660. doi: 10.1111/bjh.16424. Epub 2020 Mar 16. PMID 32180219
- [Background] Zinzani PL, Mayer J, Flowers CR, Bijou F, De Oliveira AC, Song Y, Zhang Q, Merli M, Bouabdallah K, Ganly P, Zhang H, Johnson R, Martin Garcia-Sancho A, Provencio Pulla M, Trneny M, Yuen S, Tilly H, Kingsley E, Tumyan G, Assouline SE, Auer R, Ivanova E, Kim P, Huang S, Delarue R, Trotman J. ROSEWOOD: A Phase II Randomized Study of Zanubrutinib Plus Obinutuzumab Versus Obinutuzumab Monotherapy in Patients With Relapsed or Refractory Follicular Lymphoma. J Clin Oncol. 2023 Nov 20;41(33):5107-5117. doi: 10.1200/JCO.23.00775. Epub 2023 Jul 28. PMID 37506346
- [Background] Zinzani PL, Munoz J, Trotman J. Current and future therapies for follicular lymphoma. Exp Hematol Oncol. 2024 Aug 22;13(1):87. doi: 10.1186/s40164-024-00551-1. PMID 39175100
- [Background] Morschhauser F, Fowler NH, Feugier P, Bouabdallah R, Tilly H, Palomba ML, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Daguindau N, Le Gouill S, Pica GM, Martin Garcia-Sancho A, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Zachee P, Sehn LH, Tobinai K, Cartron G, Liu D, Wang J, Xerri L, Salles GA; RELEVANCE Trial Investigators. Rituximab plus Lenalidomide in Advanced Untreated Follicular Lymphoma. N Engl J Med. 2018 Sep 6;379(10):934-947. doi: 10.1056/NEJMoa1805104. PMID 30184451
- [Background] Pott C, Jurinovic V, Trotman J, Kehden B, Unterhalt M, Herold M, Jagt RV, Janssens A, Kneba M, Mayer J, Young M, Schmidt C, Knapp A, Nielsen T, Brown H, Spielewoy N, Harbron C, Bottos A, Mundt K, Marcus R, Hiddemann W, Hoster E. Minimal Residual Disease Status Predicts Outcome in Patients With Previously Untreated Follicular Lymphoma: A Prospective Analysis of the Phase III GALLIUM Study. J Clin Oncol. 2024 Feb 10;42(5):550-561. doi: 10.1200/JCO.23.00838. Epub 2023 Dec 14. PMID 38096461
- [Background] Marcus R, Davies A, Ando K, Klapper W, Opat S, Owen C, Phillips E, Sangha R, Schlag R, Seymour JF, Townsend W, Trneny M, Wenger M, Fingerle-Rowson G, Rufibach K, Moore T, Herold M, Hiddemann W. Obinutuzumab for the First-Line Treatment of Follicular Lymphoma. N Engl J Med. 2017 Oct 5;377(14):1331-1344. doi: 10.1056/NEJMoa1614598. PMID 28976863
- [Background] Casulo C, Byrtek M, Dawson KL, Zhou X, Farber CM, Flowers CR, Hainsworth JD, Maurer MJ, Cerhan JR, Link BK, Zelenetz AD, Friedberg JW. Early Relapse of Follicular Lymphoma After Rituximab Plus Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone Defines Patients at High Risk for Death: An Analysis From the National LymphoCare Study. J Clin Oncol. 2015 Aug 10;33(23):2516-22. doi: 10.1200/JCO.2014.59.7534. Epub 2015 Jun 29. PMID 26124482
- [Background] Freedman A, Jacobsen E. Follicular lymphoma: 2020 update on diagnosis and management. Am J Hematol. 2020 Mar;95(3):316-327. doi: 10.1002/ajh.25696. Epub 2019 Dec 22. PMID 31814159